CLINICAL TRIAL: NCT06330493
Title: Prospective Multi-Center Randomized Controlled Trial to Evaluate the Safety and Efficacy of AcoArt Litos Paclitaxel Coated Percutaneous Transluminal Angioplasty (PTA) Balloon Versus Non-Coated Standard Balloon Angioplasty for the Treatment of Infrapopliteal Obstructions in Patients With Chronic Limb-Threatening Ischemia
Brief Title: AcoArt Litos PCB Below-the-knee Global Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AcoArt BTK Global Trial
Record Dates: First submitted 2024-03-10; First posted 2024-03-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PCB Group (Experimental): use PCB catheter(trade name: AcoArt Litos) to treat the stenosis or occlusion in infrapopliteal artery of experimental arm
  Interventions: Device: PCB
- PTA Group (Active Comparator): use standard PTA balloon catheter to treat stenosis or occlusion in infrapopliteal artery of control group
  Interventions: Device: PTA

INTERVENTIONS:
Device: PCB — Paclitaxel coated PTA balloon catheter
  Other Names: AcoArt Litos PCB
  Arms: PCB Group
Device: PTA — Non-coated FDA cleared (US) or CE-marked (EU) standard percutaneous transluminal angioplasty balloon catheter
  Arms: PTA Group

SUMMARY:
The objective of this study is to assess whether efficacy of the AcoArt Litos PCB is superior and whether safety of AcoArt Litos PCB is noninferior to the control device (FDA cleared PTA Balloon Catheter) regarding treatment of obstructions in the infrapopliteal arteries (located distal to the P3 segment of the popliteal artery and extending to the tibiotalar joint) in patients presenting with chronic limb-threatening ischemia (CLTI)(Rutherford 4-5)

ELIGIBILITY:
Inclusion Criteria:

- General Inclusion Criteria

1. Age ≥ 18 years at the time of consent;
2. Subjects has been informed of the nature of the study, is willing to comply with all required follow-up evaluations within the defined follow-up visit windows and has signed an Institutional Review Board(IRB)/Ethics Commitee(EC) approved consent form;
3. Female subjects of childbearing potential have a negative pregnancy test ≤ 7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation. Female subjects will be exempted from this requirement in case they are sterile, infertile, or have been post-menopausal for at least 12 months (no menses);
4. Life expectancy > 1 year in the Investigator's opinion;
5. Subject presenting with documented chronic limb-threatening ischemia(CLTI) in the target limb defined as Rutherford category 4 or 5;
6. In case of Rutherford category 5: Subjects with documented wound score 0-1, infection grade 0-2 and ischemia grade 2-3 according to the wound ischemia foot infection (WIfI) classification;
7. No other prior surgical or vascular interventions within 2 weeks before and/or planned 30 days after the protocol treatment.

   * Angiographic Inclusion Criteria
8. Reference Vessel Diameter(RVD) ≥2.0 and ≤ 4.0mm and able to be treated with available device size matrix;
9. Total length of target lesion (including significant stenosis 70~99% or occlusion) ≤ 190mm;
10. The lesion must be located in the infrapopliteal arteries and above the ankle joint. Lesions may not extend proximal to the P3 segment of the popliteal artery indicated by the tibial plateau or below the tibiotalar joint(arteries of the foot). The treatment(investigational device or PTA, including pre-dilatation) may not extend beyond these indicated regions for more than 1cm;
11. Presence of documented run-off to the foot(clearly visible at least one of the following run-off vessels; dorsalis pedis or pedal arch or plantar arteries by angiography). The target vessels should give direct or indirect run-off to the foot;
12. Absence of flow-limiting(≥ 50% stenosis) in-flow lesions confirmed by angiography. Patients with flow-limiting inflow lesions can be included if the lesion(s) have been treated successfully before enrollment, with a maximum residual restenosis of ≤30% per visual assessment. If an inflow lesion must be treated within or proximal to the P3 segment of the popliteal artery, there must be a minimum of 3 cm healthy vascular segment between this(treated) lesion and the infrapopliteal target lesion;
13. Successful pre-dilatation of the(entire) target lesion. Success being documented by angiographic visual estimate of ≤ 50% residual diameter stenosis of the target lesion and no flow limiting dissection(< Grade D dissection). Target lesion is not considered non-dilatable by the operator due to concentric, circumferential calcium and target lesion can be treated successfully by balloon angioplasty without the need for bail-out stenting.

Exclusion Criteria:

- General Exclusion Criteria

1. Planned index limb amputation above the metatarsal level, or any other planned major surgery within 30 days pre- or post-procedure. A planed amputation including and below the metatarsal level(1 or multiple rays) is accepted.
2. Recent MI or stroke < 30 days prior to the index procedure;
3. Known or suspected active infection at the time of the index procedure(abnormal white blood cell count, fever, sepsis, or positive blood culture), with the exception of a localized, controlled infection of a lower extremity wound on the target limb(only WIfI infection grade 0-2 allowed);
4. Subjects with infection grade 3 and ischemia grade 0 and 1 according to WIfI classification;
5. Subjects not independently ambulating.
6. Subjects with neurotrophic ulcers, heel pressure ulcers or calcaneal ulcers with a risk for major amputation; Subjects with uncomplicated ulcers can be included;
7. Subjects with documented active osteomyelitis, excluding the phalanges, that is beyond cortical involvement of the bone per clinical judgement;
8. Subjects with vasculitis, systemic Lupus Erythematosus or polymyalgia rheumatica on active treatment;
9. Subjects with impaired renal function defined as eGFR <30 ml/min or on dialysis;
10. Patient receiving systemic corticosyeroid therapy(expected dosage exceeding 5 mg of prednisolone or equivalent, per day, during the initial 9 months after procedure);
11. Known allergies or sensitivities to heparin, aspirin(ASA), other anticoagulant/anti-platelet therapies which could not be substitued, and/or paclitaxel or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure;
12. Subjects currently enrolled in another investigational device, drug, or biological trial;
13. Femal subjects who are breast feeding at the time of enrollment;
14. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy;
15. Any severe medical comorbidities(e.g., untreated CAD/CHF, NYHA class IV heart failure, Left Ventricular ejection fraction(LVEF) </= 30%(obtained within 1 month of index procedure), severe COPD, metastatic malignacy, etc.) that would preclude compliance with the study protocol or currently receiving immune-suppressive, chemotherapeutic, or radiation therapy;

    * Angiographic Exclusion Criteria
16. Occlusions located or extending distal to the ankle joint space;
17. Untreated (≥50% measured by angiography) inflow lesion or occlusion in the ipsilateral iliac, SFA nad popliteal arteries;
18. Failure to obtain a ≤30% residual stenosis in pre-existing, hemodynamically significant(≥50% measured by angiography) in flow lesions in the ipsilateral iliac, SFA and popliteal artery. Inflow lesions should be treated per standard of care;
19. Prior stent(s) or bypass surgery within the target vessel(s) (including stents placed within target vessels during the index procedure prior to randomization);
20. Previous procedure with drug-coated balloons in the target vessels within 6 months prior to index procedure.
21. Aneurysm in the target vessel;
22. Angiographic evidence of thrombus within target limb;
23. Pre-dilatation resulted in a major(≥ Grade D) flow-limiting dissection(observed on 2 orthogonal views) or residual stenosis >50%;
24. Use of alternative therapy, e.g. atherectomy, scoring balloon, laser, radiation therapy, stents as part of target vessel treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Composite of freedom from major amputation and primary patency | 12 months
  Composite of freedom from major amputation (above ankle amputation) and primary patency at 6 months. Primary patency is defined as absence of target lesion occlusion (no flow) and/or target lesion binary restenosis as determined by duplex ultrasound or angiography and/or clinically driven target lesion revascularization (CD-TLR).
  Binary restenosis is defined as the presence of target lesion with a hemodynamically significant restenosis ≥ 50% by angiography or PSVR ≥ 2.4 by duplex ultrasound.
  CD-TLR is defined as revascularization due to restenosis of ≥ 70% in the target lesion and
  * Wound persistence and/or;
  * Increase in size of pre-existing wounds and/or;
  * Occurrence of new wounds and/or;
  * Deterioration of Rutherford Class;
  * Hemodynamic change: decrease in TBI of 0.15 or more.
Primary Safety Endpoint: Composite of MALE and POD (Major Adverse Limb Event + Peri-Operative Death) | 30 days
  Major adverse limb event (MALE, defined as the composite of above-ankle amputation or major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of the index limb involving a below-the-knee artery) and perioperative death (POD) at 30 days.

SECONDARY OUTCOMES:
Powered Secondary Endpoint: Freedom from clinically driven TLR (CD-TLR) at 12 months | 12 months
  Composite of Limb Salvage and Primary Patency includes freedom from: above ankle amputation in index limb, 100% total occlusion of target vessel, binary restenosis of target lesion and clinically-driven target lesion revascularization (CD-TLR)
Composite of Limb salvage and primary patency | 1, 3, 12, 24 and 36 months
  Composite of limb salvage and primary patency at 1, 3, 12, 24 and 36 months
Patency rate | 1, 3, 6, 12, 24, 36 months
  Patency rate is defined as the absence of target lesion occlusion(flow/no flow) as determined by duplex ultrasound and/or angiography and freedom from clinically-driven TLR;
Freedom from CD-TLR | 1, 3, 6, 12, 24, 36 months
  CD-TLR is defined as revascularization due to restenosis of ≥ 70 % in the target lesion and
  * Wound persistence and/or;
  * Increase in size of pre-existing wounds and/or;
  * Occurrence of new wounds and/or;
  * Deterioration of Rutherford Class;
  * Hemodynamic change: decrease in TBI of 0.15 or more.
Re-occlusion rate of target lesion | 1, 3, 6, 12, 24, 36 months
  Re-occlusion rate of target lesion as determined by duplex ultrasound(no flow) and/or angiography;
Rate of Major adverse events(MAE) | 1, 3, 6, 12, 24, 36 months
  MAE is defined as all-cause death, target limb major amputation and CD-TLR;
Rate of target limb major amputation | 1, 3, 6, 12, 24, 36, 48, 60 months
  Rate of target lmb major amputations at 1, 3, 6, 12, 24, 36, 48 and 60 months;
Rate of all-cause death | 1, 3, 6, 12, 24, 36, 48, 60 months
  Rate of all-cause death at 1, 3, 6, 12, 24, 36, 48 and 60 months;
Amputation free survival rate | 1, 3, 6, 12, 24, 36, 48, 60 months
  Amputation free survival rate at 1, 3, 6, 12, 24, 36, 48 and 60 months;
Change in ankle-brachial index(ABI) | 1, 3, 6, 12, 24, 36 months
  Change in ABI from pre-procedure to 1, 3, 6, 12, 24 and 36 months
Change in toe-brachial index(TBI) | 1, 3, 6, 12, 24 months
  Change in TBI from pre-procedure to 1, 3, 6, 12 and 24 months
Change in Rutherford category | 1, 3, 6, 12, 24 and 36 months
  Change in Rutherford category from pre-procedure to 1, 3, 6, 12, 24 and 36 months
Change in EQ-5D | 1, 3, 6, 12, 24 and 36 months
  Change in EQ-5D from pre-procedure to 1,3, 6,12, 24 and 36 months
Change in VascuQol | 1, 3, 6, 12, 24 and 36 months
  Change in VascuQol from pre-procedure to 1,3, 6,12, 24 and 36 months
Primary sustained clinical improvement | 1 year
  An improvement shift in the Rutherford classification of 1 class in amputation-free, clinically driven TLR-free surviving patients at 1 year
Secondary sustained clinical improvement | 1 year
  An improvement shift in the Rutherford classification of 1 class including the need for clinically driven TLR in amputation-free surviving patients at 1 year
Wound healing | 1, 3, 6, 12, 24 and 36 months
  The wound will be evaluated at 1, 3, 6, 12, 24 and 36months
Rate of Device Success | During the procedure(After using the PCB catheter)
  Device Success is defined as, a per device basis, the achievement of successful delivery and deployment of the study device(s) at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the delivery catheter
Rate of Technical Success | During the procedure(After using the PCB catheter)
  Technical Success is defined as successful vascular access and completion of the endovascular procedure and immediate morphological success with ≤ 50% residual diameter stenosis in the treated lesion on completion angiography
Rate of Procedure Success | within 72 hours of the index procedure
  Evidence of both acute technical success and absence of safety events(e.g., death, stroke, myocardial infraction, acute onset of limb ischemia, index bypass graft or treated segment thrombosis, and/or need for urgent/emergent vascular surgery) within 72 hours of the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schneider, MD, PhD, Principal Investigator — University of California, San Francisco; Sahil Parikh, MD, PhD, Principal Investigator — Columbia University; Thomas Zeller, MD, PhD, Principal Investigator — University of Herzzentrum Freiburg
Locations (10):
- United States (8):
  - Miami Vascular Center, Hialeah, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Columbia University/NYPH, New York, New York
  - South Charlotte General & Vascular Surgery, Charlotte, North Carolina
  - Miriam Hospital, Providence, Rhode Island
  - Clements University Hospital (UTSW), Dallas, Texas
  - Sunrise Vascular, Danville, Virginia
- Medical University Graz, Graz, Austria
- AZ Sint Blasius Hospital, Dendermonde, Belgium